CLINICAL TRIAL: NCT07233460
Title: Effect of Use of Bitter Melon, Blueberry and Cranberry as Complementary Therapy on HbA1c and Diabetes Symptom Level in Individuals With Type 2 Diabetes Mellitus: Single-blind Randomized Controlled Study
Brief Title: Effect of Using Bitter Melon, Blueberries and Cranberries on HbA1c and Diabetes Symptom Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Demirağ, Ph.D (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Sponsor-Investigator, Hatice Demirağ, Ph.D, Assistant Professor, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCS05022024
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus; Symptoms and Signs; Patient
Keywords: Type 2 Diabetes Mellitus; Complementary and alternative medicine; Symptoms and Signs; Cranberry; Bitter melon; Blueberry.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: As no reference could be made to any previous four-group study on the subject, and considering the small size of the city where the research would be conducted, it was decided to include a total of 120 individuals with T2DM in the study sample, with 30 individuals in each group (bitter melon group, blueberry group, cranberry group, and control group). However, considering reasons such as death, withdrawal from the study, or missing data, it was decided to increase the sample size by 10% to 132 individuals.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher who collected the data and the person who performed the statistics were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bitter melon Group (Experimental): Before starting the study (pre-test/week 0), all group participants first completed the "Patient Information Form" and the "Diabetes Symptom Checklist Scale," and their HbA1c venous blood values were measured. At the end of the study (post-test/12th week), the "Diabetes Symptom Checklist Scale" was administered again to individuals in the three groups, and their HbA1c venous blood values were measured. In addition, telephone follow-up was conducted to determine whether the individuals had used the powdered extracts completely for 12 weeks.
  Interventions: Other: Bitter Melon Group
- Blueberry Group (Experimental): Before starting the study (pre-test/week 0), all group participants first completed the "Patient Information Form" and the "Diabetes Symptom Checklist Scale," and their HbA1c venous blood values were measured. At the end of the study (post-test/12th week), the "Diabetes Symptom Checklist Scale" was administered again to individuals in the three groups, and their HbA1c venous blood values were measured. In addition, telephone follow-up was conducted to determine whether the individuals had used the powdered extracts completely for 12 weeks.
  Interventions: Other: Blueberry Group
- Cranberry Group (Experimental): Before starting the study (pre-test/week 0), all group participants first completed the "Patient Information Form" and the "Diabetes Symptom Checklist Scale," and their HbA1c venous blood values were measured. At the end of the study (post-test/12th week), the "Diabetes Symptom Checklist Scale" was administered again to individuals in the three groups, and their HbA1c venous blood values were measured. In addition, telephone follow-up was conducted to determine whether the individuals had used the powdered extracts completely for 12 weeks.
  Interventions: Other: Cranberry Group
- Control Group (No Intervention): Before starting the study (pre-test/week 0), all group participants first completed the "Patient Information Form" and the "Diabetes Symptom Checklist Scale," and their HbA1c venous blood values were measured. At the end of the study (post-test/12th week), the "Diabetes Symptom Checklist Scale" was administered again to individuals in the three groups, and their HbA1c venous blood values were measured.

INTERVENTIONS:
Other: Bitter Melon Group — Patients who voluntarily used bitter melon powder extract continued to consume 1 teaspoon (10 g total) of powdered extract mixed with yogurt or water twice a day (morning and evening) for 12 weeks.
  Arms: Bitter melon Group
Other: Blueberry Group — Patients who voluntarily used bitter blueberry powder extract continued to consume 1 teaspoon (10 g total) of powdered extract mixed with yogurt or water twice a day (morning and evening) for 12 weeks.
  Arms: Blueberry Group
Other: Cranberry Group — Patients who voluntarily used cranberry powder extract continued to consume 1 teaspoon (10 g total) of powdered extract mixed with yogurt or water twice a day (morning and evening) for 12 weeks.
  Arms: Cranberry Group

SUMMARY:
This double-blind, randomized controlled trial investigated the effect of bitter melon, blueberry, and cranberry powder extract use on glycemic control and diabetes symptom levels in individuals with T2DM.

DETAILED DESCRIPTION:
The increasing prevalence of Type 2 Diabetes Mellitus (T2DM) worldwide and the search for additional support to current treatments have increased interest in researching natural components such as bitter melon, blueberry, and cranberry, known for their antioxidant and hypoglycemic potential, as complementary therapies. This double-blind, randomized controlled trial investigated the effect of bitter melon, blueberry, and cranberry powder extract use on glycemic control and diabetes symptom levels in individuals with T2DM.

The study, conducted with four groups (bitter melon, blueberry, cranberry, and control), included 120 individuals diagnosed with T2DM. Individuals in the experimental group used 10g of powdered extract daily for 12 weeks, while those in the control group used nothing. The 'Patient Information Form' and 'Diabetes Symptoms Checklist Scale' were administered before the start of the study (pre-test/week 0) and at the end (post-test/week 12), and the venous blood value of the Hemoglobin A1c test (HbA1c) was measured.

In the experimental groups (bitter melon, blueberry, cranberry), after 12 weeks of treatment, statistically significant decreases were observed in HbA1c, the total score and all Subdimensions scores of the 'Diabetes Symptoms Checklist Scale', weight, and BMI compared to the control group; while in the control group, there was a significant increase in all parameters except HbA1c (p<0.05). Although there was no difference between the experimental (bitter melon, blueberry, cranberry) groups in the intergroup measurements, HbA1c, the total mean scores of the Diabetes Symptom Checklist Scale, weight, and BMI were found to be significantly lower than in the control group (p<0.05).

Bitter melon, blueberry, and cranberry powder extracts were found to be equally effective in reducing HbA1c, diabetes symptoms, weight, and BMI in T2DM patients. The lack of difference in efficacy between the three extracts in terms of glycemic and symptom levels suggests that these three natural products can be considered equivalent therapeutic options in the complementary treatment of T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Volunteering to participate in the study,
* Being conscious and able to communicate,
* Having been diagnosed with T2DM at least 3 months prior and currently using oral antidiabetic medication,
* Be using one of the following powder extracts-bitter melon, blueberry, or cranberry-for the first time as a complementary treatment upon a physician's recommendation and be on the first day of use,
* Not taking any other medications that affect blood sugar,
* No allergy to bitter melon, blueberry, or cranberry,
* Not engaging in exercise,
* Taking 10g of bitter melon, blueberry, or cranberry powder extract daily.

Exclusion Criteria:

* Not meeting the inclusion criteria, having a known psychological disorder,
* Having previously received complementary therapy for DM, or having hearing loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 week
  Unlike instant blood glucose values, HbA1c reliably reflects an individual's average blood sugar level over the past two to three months by measuring the amount of glucose bound to hemoglobin during the average lifespan of erythrocytes (approximately 120 days).
  Before starting the study (pre-test/week 0) HbA1c venous blood values were measured. Patients who voluntarily used bitter melon, blueberry, or cranberry continued to consume 1 teaspoon (10 g total) of powdered extract mixed with yogurt or water twice a day (morning and evening) for 12 weeks. At the end of the study (post-test/12th week), the was administered again to individuals HbA1c venous blood values were measured.
Diabetes Symptom Checklist Scale | 12 week
  The scale consists of a total of 34 items. These categories are: neurology (3, 11, 15, 21, 25, 34), psychology (1, 2, 4, 6, 17, 20), cardiology (5, 8, 9, 13, 24, 26, 29, 30), ophthalmology (10, 14, 22, 28), psychology/cognition (7, 19, 27, 31, 33), and hyperglycemia (12, 16, 23, 32) Subdimensionss. Responses on the scale are numbered from 0 to 5, with "0" meaning "none" and "5" meaning "extremely."
  Before starting the study (pre-test/week 0), all group participants first completed "Diabetes Symptom Checklist Scale" were measured. Patients who voluntarily used bitter melon, blueberry, or cranberry continued to consume 1 teaspoon (10 g total) of powdered extract mixed with yogurt or water twice a day (morning and evening) for 12 weeks. At the end of the study (post-test/12th week), the "Diabetes Symptom Checklist Scale" was administered again to individuals were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Demirağ, Principal Investigator — Study Principal Investigator Gümüşhane Universıty
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Maybe I will decide later.